CLINICAL TRIAL: NCT02180399
Title: Role of the Serial Measurement of Capillary Blood Lactate in the Management of Sepsis Outside the Intensive Care
Brief Title: Serial Measurement of Capillary Blood Lactate in the Management of Sepsis
Acronym: SepsisMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6031
Record Dates: First submitted 2014-02-05; First posted 2014-07-02 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
Keywords: Sepsis; Capillary blood lactate; Serial measurement of capillary
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Determination of capillary lactate by using "point-of-care" technique is accessible, fast and allows to quantify the circulatory and metabolic dysfunction caused by sepsis. Compared to conventional assay techniques in arterial blood, capillary assay technique may have an increased susceptibility to metabolic alterations induced by sepsis in its initial stages. This increased sensitivity is not necessarily relevant in the management of the most serious patients for whom the diagnosis is obvious, but it could be very useful in patients for whom a diagnosis of severe sepsis or shock have not yet been adopted, particularly to help better identify patients who would require intensive management and avoid the installation of these serious disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Installation without any plausible explanation of at least one of the following clinical criteria:

  * Chills, fever, mottling, respiratory rate> 20/min; Sat02 < 90% or > 94% with more than 4l O2, heart rate > 90/min,systolic blood pressure < 100 mmHg or 40 mmHg lower compared with normal values, Glasgow coma score < 14. or: .a combination of two (or more) of clinical and laboratory criteria for sepsis.
* Signed informed consent form

Exclusion Criteria:

* Need in its current treatment of aerosol administration of beta agonists at a frequency greater than one per 8 hours;
* Targeted therapeutic measures have already stated for more than 60 minutes;
* Diagnosis other than Sepsis;
* Malignant neoplasm or other progressive disease and expected survival was less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over age 18 with an acute systemic inflammatory response syndrome array of presumed infectious not yet been treated.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
measurement of capillary blood lactate | 72 hours after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ANDRES, MD, PhD, Study Director — University Hospitals of Strasbourg
Locations (2):
- France (2):
  - SERVICE DE MED. INTERNE - DIABETE ET MALADIES METABOLIQUES, 1-place de l'Hôpital, Strasbourg
  - Service de Médecine Interne - Clinique Médicale B, Strasbourg